CLINICAL TRIAL: NCT05371821
Title: Cardiac Assessment of Obese and Overweight Children Attending Asyut University Children Hospital
Brief Title: Cardiac Assessment in Obese and Overweight Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Osman Gamal Hassan, Cardiac assessment of obese and overweight children attending Asyut University children hospital, Assiut University
Other Study IDs: assessment of obese children
Record Dates: First submitted 2022-04-23; First posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Echocardiography — Echocardiographic parameters in obese and overweight

SUMMARY:
Is to assess cardiac functions of overweight and obese children attending assiut University children hospital in one year duration .

DETAILED DESCRIPTION:
The prevalence of overweight and obesity in children is increasing worldwide at an alarming rate in both developing and developed countries .the relation between obesity and cardiac structure and function in children is less well documented and conflicting results have been reported .In addition, obesity is associated with a heterogeneity of metabolic abnormalities , (e.g., dyslipidemia , insulin resistance hyperglycaemia and hypertension , that may provide a plausible biologic link between obesity and the increased risk of cardiovascular morbidity and mortality .The clustering of these risk factors for cardiovascular disease is referred to as the "metabolic syndrome." Although the concept and definition of the metabolic syndrome are controversial at the moment, there is no doubt that a cluster of cardiovascular risk factors is present in obese children and adolescents and that their presence increases with worsening obesity .children are likely to be the ideal candidates for providing insight into the myocardial changes related to obesity because they are suggested to be free of other cardiovascular risk factors indifferent echocardiographic studies .

ELIGIBILITY:
Inclusion Criteria:

1. - Age: children at 2-18 years .
2. - Overweight children whose body mass index at or above the 85th percentile and below the 95th percentile for the same age and sex
3. - Obese children whose body mass index at or above the 95th percentile for the same age and sex.

Exclusion Criteria:

1- Obese children below two years 2 - Cases with syndromic obesity, diabetes

* thyroid and parathyroid and those with congenital heart diseases

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Obese and overweight children from 2 years till age of 18 years .
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-05-20 (Estimated); Primary Completion 2023-04-21 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Cardiac assessment of obese and overweight children | Baseline
  Echocardiography performed by an expert cardiologist using a Philips envisor c machine to assess the following parameters (left ventricle end-diastolic diameter (LVEDD), left ventricle end-systolic diameter (LVESD), interventricular septal systolic diameter (IVSSD), interventricular septal diastolic diameter (IVSDD) left ventricle fraction shortening (FS), left ventricle ejection fraction (EF), left atrium to aorta ratio (LA:AO), mitral annular plane area systolic excursion (MAPSE), fraction area shortening of the right ventricle (FAC), tricuspid annular plane systolic excursion (TAPSE)
Assessment of body mass index | baseline
  BMI described in kg / m²

REFERENCES:
- [Result] Bates JH, Serdula MK, Khan LK, Jones DA, Macera CA, Ainsworth BE. Intensity of physical activity and risk of coronary heart disease. JAMA. 2001 Jun 20;285(23):2973; author reply 2974. No abstract available. PMID 11410086
- [Result] de Simone G, Daniels SR, Devereux RB, Meyer RA, Roman MJ, de Divitiis O, Alderman MH. Left ventricular mass and body size in normotensive children and adults: assessment of allometric relations and impact of overweight. J Am Coll Cardiol. 1992 Nov 1;20(5):1251-60. doi: 10.1016/0735-1097(92)90385-z. PMID 1401629
- [Result] Kono Y, Yoshinaga M, Oku S, Nomura Y, Nakamura M, Aihoshi S. Effect of obesity on echocardiographic parameters in children. Int J Cardiol. 1994 Aug;46(1):7-13. doi: 10.1016/0167-5273(94)90111-2. PMID 7960279
- [Result] Yoshinaga M, Yuasa Y, Hatano H, Kono Y, Nomura Y, Oku S, Nakamura M, Kanekura S, Otsubo K, Akiba S, et al. Effect of total adipose weight and systemic hypertension on left ventricular mass in children. Am J Cardiol. 1995 Oct 15;76(11):785-7. doi: 10.1016/s0002-9149(99)80227-6. PMID 7572655
- [Result] Daniels SR, Kimball TR, Morrison JA, Khoury P, Witt S, Meyer RA. Effect of lean body mass, fat mass, blood pressure, and sexual maturation on left ventricular mass in children and adolescents. Statistical, biological, and clinical significance. Circulation. 1995 Dec 1;92(11):3249-54. doi: 10.1161/01.cir.92.11.3249. PMID 7586311
- [Result] Goran MI, Gower BA. Abdominal obesity and cardiovascular risk in children. Coron Artery Dis. 1998;9(8):483-7. doi: 10.1097/00019501-199809080-00003. No abstract available. PMID 9847979
- [Result] Steinberger J, Daniels SR; American Heart Association Atherosclerosis, Hypertension, and Obesity in the Young Committee (Council on Cardiovascular Disease in the Young); American Heart Association Diabetes Committee (Council on Nutrition, Physical Activity, and Metabolism). Obesity, insulin resistance, diabetes, and cardiovascular risk in children: an American Heart Association scientific statement from the Atherosclerosis, Hypertension, and Obesity in the Young Committee (Council on Cardiovascular Disease in the Young) and the Diabetes Committee (Council on Nutrition, Physical Activity, and Metabolism). Circulation. 2003 Mar 18;107(10):1448-53. doi: 10.1161/01.cir.0000060923.07573.f2. No abstract available. PMID 12642369
- [Result] Aggoun Y. Obesity, metabolic syndrome, and cardiovascular disease. Pediatr Res. 2007 Jun;61(6):653-9. doi: 10.1203/pdr.0b013e31805d8a8c. PMID 17426660
- [Result] Weiss R, Dziura J, Burgert TS, Tamborlane WV, Taksali SE, Yeckel CW, Allen K, Lopes M, Savoye M, Morrison J, Sherwin RS, Caprio S. Obesity and the metabolic syndrome in children and adolescents. N Engl J Med. 2004 Jun 3;350(23):2362-74. doi: 10.1056/NEJMoa031049. PMID 15175438
- [Result] Di Salvo G, Pacileo G, Del Giudice EM, Natale F, Limongelli G, Verrengia M, Rea A, Fratta F, Castaldi B, D'Andrea A, Calabro P, Miele T, Coppola F, Russo MG, Caso P, Perrone L, Calabro R. Abnormal myocardial deformation properties in obese, non-hypertensive children: an ambulatory blood pressure monitoring, standard echocardiographic, and strain rate imaging study. Eur Heart J. 2006 Nov;27(22):2689-95. doi: 10.1093/eurheartj/ehl163. Epub 2006 Aug 11. PMID 16905554
- [Result] Labombarda F, Zangl E, Dugue AE, Bougle D, Pellissier A, Ribault V, Maragnes P, Milliez P, Saloux E. Alterations of left ventricular myocardial strain in obese children. Eur Heart J Cardiovasc Imaging. 2013 Jul;14(7):668-76. doi: 10.1093/ehjci/jes238. Epub 2012 Nov 15. PMID 23161790
- [Result] Li X, Li S, Ulusoy E, Chen W, Srinivasan SR, Berenson GS. Childhood adiposity as a predictor of cardiac mass in adulthood: the Bogalusa Heart Study. Circulation. 2004 Nov 30;110(22):3488-92. doi: 10.1161/01.CIR.0000149713.48317.27. Epub 2004 Nov 22. PMID 15557363